CLINICAL TRIAL: NCT06683898
Title: The Role of Focus Strategies on Pilates Performance and Reaction Time: A Randomized Controlled Trial
Brief Title: The Role of Focus Strategies on Pilates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, Asistant Professor, Physiotherapist, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09.11.2024
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Reaction Time; Humans; Exercise Therapy; Exercise Movement Techniques; Pilates

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Focused Pilates (Experimental): Pilates training was implemented with an external focus (EF).
  Interventions: Other: External Focused Pilates; Other: Internal Focused Pilates
- Internal Focused Pilates (Experimental): Pilates training was implemented with an internal focus (IF).
  Interventions: Other: External Focused Pilates; Other: Internal Focused Pilates

INTERVENTIONS:
Other: External Focused Pilates — Pilates training was implemented with an external focus (EF).
Other: Internal Focused Pilates — Pilates training was implemented with an internal focus (IF).

SUMMARY:
Aims of the randomized controlled study is compare to the effects of external and internal focus strategies, commonly used in Pilates, on participants' reaction time and performance metrics. Conducted over an 8-week Pilates program at Alanya Alaaddin Keykubat University, we plan to include 25 participants in each focus group. Participants in the external focus group will use equipment to perform exercises, while the internal focus group will perform exercises with attention to body positioning.

DETAILED DESCRIPTION:
The primary aim of this study is to examine the difference in effects between 8-week internally and externally focused Pilates exercises on the performance of young sedentary individuals. A secondary aim is to investigate the effects of internally and externally focused Pilates exercises on the physical characteristics and reaction time of young sedentary individuals.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged between 18 and 30 years who have no musculoskeletal disabilities and are willing to exercise were included in the study.

Exclusion Criteria:

* Had any cardiovascular or musculoskeletal condition that would prevent them from exercising,
* Had an acute pain history of 5 or more on the visual analog scale in the past week,
* Had a systemic disease that would prevent exercise,
* Had a BMI of 30 or above,
* Had any issues that would hinder their ability to perceive or understand verbal commands, or had hearing problems.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-10-05 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Multiple Jump Test | Baseline - right after the intervention
  15-Second Continuous Jump Test
BFS Vertical Jump Test | Baseline - right after the intervention
  The Vertical Jump Test is a practical test that provides information about an individual's anaerobic power level.
Squat Jump Test | Baseline - right after the intervention
  The explosive strength characteristic demonstrated by the leg muscles is measured based on their maximal force.
Acoustic Reaction Test | Baseline - right after the intervention
  This test measures the time between a visual/auditory stimulus and the athlete's response movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Alaaddin Keykubat Üniversity, Antalya, Alanya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No